CLINICAL TRIAL: NCT02094378
Title: A Randomized, Double-blind, Placebo-controlled, 2-period Crossover Study to Evaluate the Effect of Intranasal Esketamine on Cognitive Functioning in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Intranasal Esketamine on Cognitive Functioning in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CR103823; ESKETINTRD1005 (Other: Janssen Research & Development, LLC); 2014-000468-16 (EudraCT Number)
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Healthy; Esketamine; Cognitive functioning
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esketamine-Placebo (Experimental): Participants assigned to treatment sequence 1 will receive 84 mg esketamine intranasally on Day 1 of Period 1 and then receive placebo intranasally on Day 1 in Period 2. Periods 1 and 2 will be separated by 7 days.
  Interventions: Drug: Esketamine; Drug: Placebo
- Placebo-Esketamine (Placebo Comparator): Participants assigned to treatment sequence 2 will receive placebo intranasally on Day 1 of Period 1 and then receive 84 mg esketamine intranasally on Day 1 in Period 2. Periods 1 and 2 will be separated by 7 days.
  Interventions: Drug: Esketamine; Drug: Placebo

INTERVENTIONS:
Drug: Esketamine — 84 mg esketamine administered intranasally
Drug: Placebo — Placebo administered intranasally

SUMMARY:
The purpose of this study is to assess the cognitive effects associated with administration of intranasal esketamine 84 mg.

DETAILED DESCRIPTION:
This is a randomized (participants assigned to 1 of 2 treatment sequences by chance), double-blind (identity of study drugs will not be known to participant or members of study staff), placebo-controlled (a substance without active drug identical in appearance to esketamine), 2-period crossover study (participants assigned to each treatment sequence will receive 1 dose of esketamine and 1 dose of placebo administered intranasally [through the nose]) conducted in healthy adult participants at a single center. Participants will complete 3 study phases: A screening phase of up to 3 weeks; a 2-week double-blind treatment phase, which includes 2 treatment periods (Periods 1 and 2) separated by a washout interval of at least 7 days; and, a 1-week posttreatment (follow up) phase, if applicable. The duration of the study for each participant will be approximately 6 weeks. Blood and urine samples will be collected during the study for laboratory assessments. Participants will be monitored for safety from the time of signing the informed consent form up until 1 week after the last dose of study drug (or end of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) (weight [kg]/height[m2]) between 18 and 30 kg/m2 (inclusive), and body weight not less than 45 kg
* Blood pressure (after the subject is supine for 5 minutes) between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic at Screening and predose on Day 1 of Period 1
* A 12-lead ECG consistent with normal cardiac conduction and function at Screening and predose on Day 1 of Period 1
* Comfortable with self-administration of intranasal medication and able to follow instructions provided
* Non-smoker for at least 6 months before first study drug administration

Exclusion Criteria:

* Subject has clinically significant liver or renal insufficiency; cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances. A significant primary sleep disorder is exclusionary
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or on Day 1 of Period 1, as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12-lead ECG at screening or on Day 1 of Period 1, as deemed appropriate by the investigator
* Anatomical or medical conditions that may impede delivery or absorption of study medication (e.g., undergone facial reconstruction, rhinoplasty, significant structural or functional abnormalities of the nose or upper airway; obstructions or mucosal lesions of the nostrils or nasal passages; undergone sinus surgery in the previous 2 years; or signs and symptoms of rhinitis predose on Day 1 of Period 1)
* Has an abnormal or deviated nasal septum with any 1 or more of the following symptoms: blockage of 1 or both nostrils, nasal congestion (especially 1-sided), frequent nosebleeds, frequent sinus infections, and at times has facial pain, headaches, and postnasal drip

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cognitive functioning measured by the The Cogstate® Computerized Battery | On Day 1 at -1 hour, 40 minutes, and at 2, 4, and 6 hours after dosing (or at the end of treatment)
  The Cogstate® Computerized Battery of tests will include 5 tests: Detection (simple reaction time task measuring processing speed [lower score = better performance]); Identification (choice reaction time paradigm measuring attention [lower score = better performance]); One Card Learning (visual episodic memory measure [higher score = better performance]); One Back ( "n-back" working memory measure [higher score = better performance]); and, Groton Maze Learning Test (executive function measure; total number of errors made in attempting to learn the same hidden pathway on five consecutive trials at a single session [lower score = better performance]) (Maruff 2004, Snyder 2005).
Change from baseline in cognitive functioning measured by the Karolinska Sleepiness Scale (KSS) | On day 1 at -1 hour, 40 minutes, and at 2, 4, and 6 hours after dosing (or at the end of treatment)
  The KSS is a subject-reported assessment used to rate sleepiness on a scale of 1 to 9, ranging from 'extremely alert' (1) to 'very sleepy, great effort to keep awake, fighting sleep' (9) (Akerstedt 1990).
Change from baseline in cognitive functioning measured by the mental effort scale | On Day 1 at -1 hour, 40 minutes, and at 2, 4, and 6 hours after dosing (or at the end of treatment)
  The mental effort scale is a subject-reported assessment of the level of effort needed to complete the test battery on a 15-cm equal interval scale (Zijlstra1993).

SECONDARY OUTCOMES:
The concentration of esketamine and noresketamine from time zero to the last observable concentration (AUClast) | Day 1 at 0, 10, and 40 minutes and 1, 2, and 4 hours after dosing
The maximum plasma concentration (Cmax) of esketamine and noresketamine | Day 1 at 0,10, and 40 minutes and at 1, 2, 4, and 6 hours after dosing
Time to Maximum Plasma Concentration (Tmax) of esketamine and noresketamine | Day 1 at 0, 10, and 40 minutes and 1, 2, 4, and 6 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Leiden, Netherlands

REFERENCES:
- [Derived] Morrison RL, Fedgchin M, Singh J, Van Gerven J, Zuiker R, Lim KS, van der Ark P, Wajs E, Xi L, Zannikos P, Drevets WC. Effect of intranasal esketamine on cognitive functioning in healthy participants: a randomized, double-blind, placebo-controlled study. Psychopharmacology (Berl). 2018 Apr;235(4):1107-1119. doi: 10.1007/s00213-018-4828-5. Epub 2018 Feb 1. PMID 29392371